CLINICAL TRIAL: NCT00252434
Title: Behavioral Therapy Development for Methamphetamine Abuse
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R21DA018075 (NIH)
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Depression; Drug Abuse; Sexually Transmitted Diseases
Keywords: high-risk sexual behavior; methamphetamine use; drug craving; addiction behaviors
MeSH Terms: conditions — Depression; Substance-Related Disorders; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy Development for Methamphetamine Abuse

SUMMARY:
The purpose of this study is to evaluate whether a specially developed group counseling approach is better able to help HIV-positive gay and bisexual men (GBM) who use crystal meth to stop using methamphetamines, reduce sexual risk behaviors, and stay on their HIV medications than a standard drug treatment program. Another purpose is to determine whether having a drug abuse treatment program in an HIV medical clinic makes it easier to attend treatment than going to a separate location for drug abuse treatment.

DETAILED DESCRIPTION:
The study features activities that include development and refinement of a culturally-specific cognitive behavioral therapy that integrates aspects of drug abuse treatment with HIV medication adherence interventions and cultural elements of being a gay or bisexual man receiving medical care for HIV/AIDS. To estimate the size of the signal of this intervention, the study proposes a two parallel group design in which 50 treatment-seeking HIV-seropositive gay and bisexual men who meet criteria for methamphetamine abuse and who receive HIV medical care at the UCLA Center for Clinical AIDS Research and Education (CARE) clinic are randomized to the study condition or a treatment-as-usual (TAU) condition. Participants assigned to the experimental condition receive 12 weeks of twice-weekly GCBT, with a 6-months post-randomization follow-up visit. Participants assigned to the TAU condition are referred to the UCLA Addiction Medicine Clinic (AMC), where they receive the clinic's standard of care treatment for methamphetamine dependence for 12 weeks, and return for a 6-month follow-up visit. Analyses are conducted on all participants who meet inclusion/exclusion criteria, express desire for treatment, and receive at least one "dose" of the cognitive-behavioral treatment or make one visit to the AMC. Participants in both conditions agree to weekly and monthly data collection visits, including the provision of urine samples. Primary outcome variables are methamphetamine use, sexual risk behaviors, and HIV medication compliance. The proposed design maintains the focus on intervention development and feasibility, while recognizing that the second phase of this development will be informed by having accurate estimates of effect sizes for the intervention and adequate resources to conduct the full-scale trial.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-seropositive, GBM receiving medical treatment for HIV for at least 30 days prior to signing informed consent at the University of California, Los Angeles (UCLA) Center for Clinical AIDS Research and Education (CARE) clinic, aged 18-65
2. Willing to give informed consent and comply with study procedures
3. Willing to provide consent to contact treating physicians and pharmacies to assess adherence to HIV medications
4. Diagnosed with current methamphetamine abuse as determined by Mini-International Neuropsychiatric Interview (MINI)
5. Interested in seeking treatment for methamphetamine abuse and in participating in this research project.

Exclusion Criteria:

1. Unwilling to give, or withdrawal of, informed consent
2. Inability to understand nature of study
3. A psychiatric condition that, in the principal investigator's judgment, warrants additional intervention to ensure participant safety (e.g., meets Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision [DSM-IV-TR] criteria for current bipolar disorder or a psychotic disorder)
4. Current suicidal ideation or suicide attempt within the past 3 months
5. Concurrent dependence on opiates, alcohol, or benzodiazepines as determined by MINI.
6. Total lack of any type of healthcare coverage. These potential participants will be given low-fee treatment referrals.

Ages: 18 Years to 65 Years | Sex: Male
Age Groups: Adult, Older Adult
Dates: Start 2004-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
methamphetamine use | weekly

SECONDARY OUTCOMES:
sexual risk behaviors | monthly

CONTACTS AND LOCATIONS:
Overall Officials: James A. Peck, PsyD., Principal Investigator — UCLA Integrated Substance Abuse Programs; James A Peck, Psy.D., Principal Investigator — UCLA Integrated Substance Abuse Programs
Locations (1):
- UCLA Center for Clinical AIDS Research and Education (CARE) Clinic, Los Angeles, California, United States